CLINICAL TRIAL: NCT02208167
Title: IGHID 1320 - A Phase I Study to Evaluate the Safety, Immunologic, and Virologic Responses of HIV-1 Antigen Expanded Specific T Cell Therapy (HXTC) as a Therapeutic Strategy in HIV-Infected Individuals Started on Antiretroviral Therapy During Acute and Chronic Infection
Brief Title: Phase I Study of HIV 1 Antigen Expanded Specific T Cell Therapy
Acronym: HXTC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: CARE Collaboratory of AIDS Researchers for Eradication (Unknown); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0741; 5U19AI096113-05 (NIH)
Record Dates: First submitted 2014-07-24; First posted 2014-08-04 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2018-02

CONDITIONS: HIV
Keywords: Antigen Expanded Specific T Cell Therapy; HXTC; Antiretroviral Therapy; Acute HIV infection; Chronic HIV infection; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronic HIV infection (Other): HXTC infusion
  Interventions: Biological: HXTC infusion
- Acute HIV infection (Other): HXTC infusion
  Interventions: Biological: HXTC infusion

INTERVENTIONS:
Biological: HXTC infusion
  Other Names: HIV 1 antigen expanded specific T cell

SUMMARY:
This is a phase 1, single-site study is to evaluate the safety and immunologic and virologic efficacy of ex vivo expanded HIV-1 multi-antigen specific T-cell (HXTC) therapy in HIV-infected individuals with viral suppression on antiretroviral therapy (ART).

DETAILED DESCRIPTION:
The main hypothesis of this study is that the administration of autologous ex vivo expanded HIV-specific T-cells (HXTCs) primed to recognize multiple HIV-1 antigens in HIV-infected participants who initiated ART during acute and chronic HIV infection will be safe, increase HIV-1 antigen specific T-cell immune responses and decrease low level viremia.

In addition, secondary objectives are to:

1. Determine the feasibility of manufacturing HXTC from participants who started cART during acute and chronic HIV infection.
2. Explore the ability of autologous ex vivo expanded HIV-1 specific T-cells (HXTC) to increase HIV-1 specific immune responses in participants initiated on cART during acute and chronic HIV infection.
3. Explore the ability of autologous ex vivo expanded HIV-1 specific T-cells (HXTC) to impact latent HIV infection as measured by a quantitative viral outgrowth assay (QVOA) and integrated proviral DNA quantification, and low level viremia as measured by a single copy assay (SCA) in participants initiated on cART during acute and chronic HIV infection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years and ≤65 years of age
2. Confirmation of HIV 1 infection

   * Chronic HIV infection (CHI) is defined as documentation of a positive HIV test result by any licensed ELISA test kit and confirmed by Western blot or Multispot HIV 1/HIV 2 assay prior to screening. HIV culture, HIV antigen, plasma HIV RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
   * Acute HIV infection (AHI) is defined as: 1) a negative or indeterminate enzyme immunoassay (EIA) plus a reproducibly detectable HIV by amplification methods, or 2) a positive 4th generation HIV Ag/Ab Combination assay and either a negative/indeterminate HIV rapid test or a negative/indeterminate Western blot, or 3) a negative HIV RNA test within 45 days of a positive EIA and ART initiation.

   Note: the HIV definitions above are pertinent to the time of diagnosis and treatment initiation.
3. AHI participants are defined as HIV infected patients on suppressive ART that was initiated within 45 days of AHI diagnosis as defined in protocol section 5.1.2.
4. CHI participants are defined as HIV infected patients who initiated ART with chronic HIV as defined in protocol section 5.1.2.
5. On potent antiretroviral therapy, defined as at least 2 nucleoside/nucleotide reverse transcriptase inhibitors plus a non-nucleoside reverse transcriptase inhibitor, integrase inhibitor, or a protease inhibitor without interruption (defined as missing doses for more than two (2) consecutive days or more than four (4) cumulative days) in the 12 weeks prior to entry.

   Other potent fully suppressive antiretroviral combinations will be considered on a case by case basis. Prior changes in or elimination of medications for easier dosing schedule, intolerance, toxicity, or other reasons are permitted if an alternative suppressive regimen was maintained.
6. Stable ART regimen for minimum of 3 months. NOTE: The ART regimen is defined by current treatment guidelines. Participants may have had one or more changes in their ART regimen for tolerance, change of guidelines, or dosing simplification.
7. Ability and willingness of participant to continue cART throughout the study.
8. Plasma HIV 1 RNA below detected limit by conventional assays (limit of detection: 75, 50, 40, or 20 copies/mL) for ˃1 year.

   A single unconfirmed plasma HIV RNA ˃ limit of detection but ˂ 1000 c/mL allowed within the prior 12 months; but none in the preceding 6 months.
9. Plasma HIV 1 RNA ˂ 50 copies/mL at screening.
10. CD4+ cell count ˃ 350 cells/mm3 at screening.
11. No active HCV infection (measureable HCV RNA) within 90 days of enrollment.
12. No active HBV infection (measureable HBV DNA or HBVsAg+) within 90 days of enrollment.
13. All female participants participating in sexual activity that could lead to pregnancy must agree to use at least two of the following reliable methods of birth control (at least one of which is a barrier method) for at least 21 days prior to study entry and until 12 weeks after the last dose of the study product: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, Intrauterine Device, hormone-based contraceptive, tubal ligation, NuvaRing.
14. All male participants participating in sexual activity that could lead to pregnancy must agree to use condoms for at least 21 days prior to study entry and until 12 weeks after the last dose of the study product.
15. Ability and willingness of subject to give written informed consent.
16. Ability and willingness to provide adequate locator information.
17. Ability and willingness to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the Protocol requirements.
18. Adequate vascular access for HXTC infusion and leukapheresis.
19. Potential participant must have adequate organ function as indicated by the following laboratory values:

Absolute neutrophil count (ANC): ≥ 1,500 /mcL Platelets: ≥ 125,000 / mcL Hemoglobin: ≥ 12 g/dL

Coagulation:

Prothrombin Time or INR: ≤ 1.5 times upper limit of normal (ULN)

Chemistry K+ levels: Within normal limits

Renal:

Serum creatinine (or calculated creatinine clearance* for those with creatinine > 1.3 ULN): ≤ 1.3 times upper limit of normal (ULN); OR Creatinine clearance* ≥ 60 mL/min for potential participants with creatinine levels > 1.3 times institutional ULN

Hepatic Serum total bilirubin: Total bilirubin < 1.5 times the upper limit of the normal range. If total bilirubin is elevated, direct bilirubin must be < 2 times the ULN range.

NOTE: If participant is on an atazanavir containing therapy then a direct bilirubin should be measured instead of the total bilirubin and must be ≤ 1.0mg/dL.

AST (SGOT) and ALT (SGPT): ≤ 2.0 times ULN Alkaline Phosphatase: ≤ 2.5 times ULN

*Creatinine clearance should be calculated per institutional standard.

Exclusion Criteria:

1. Prior use of any HIV immunotherapy or vaccine within 12 months prior to Screening.
2. Use of any of the following within 90 days prior to entry: immunomodulatory, cytokine, or growth stimulating factors such as systemic corticosteroids, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, IFN, interleukin 2 (IL 2), Coumadin, warfarin, or other Coumadin derivative anticoagulants.
3. Received any infusion blood product, immune globulin, or hematopoietic growth factors within 90 days prior to study entry.
4. Pregnancy or breast-feeding.
5. History or other evidence of severe illness, malignancy, immunodeficiency other than HIV, or any other condition that would make the subject unsuitable for the study in the opinion of the investigator.
6. Use of topical steroids over a total area exceeding 0.5mg/kg/day within 30 days prior to Screening.
7. Any active malignancy that may require chemotherapy or radiation therapy.
8. Compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric illness or a physical illness, e.g., infectious disease. Prisoner recruitment and participation is not permitted.
9. Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) within 4 weeks prior to study entry.
10. Unable to have a person available to drive participant home at infusion visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Safety | 1st day of study treatment until 28 days post last infusion
  Occurrence of any ≥ Grade 3 AE including signs/symptoms, lab toxicities, and/or clinical events, that are: possibly, probably or definitely related to study treatment.

SECONDARY OUTCOMES:
Secondary Safety | 1st day of study treatment through Week 48
  Occurrence of any ≥ Grade 3 AE including signs/symptoms, lab toxicities, and/or clinical events regardless of adjudicated relationship to study treatment.

OTHER OUTCOMES:
Immune Response | baseline, weeks 1, 2, 4, 6, 8, 13, 24, 36, and 48 post-infusion
  Frequency of HIV-1 antigen-specific (gag, pol, nef) CD8+ T-cells by ELIspot
Immune Response | baseline, weeks 1, 2, 4, 6, 8, 13, 24, 36, and 48 post-infusion
  Change in T cell responses from baseline to post-infusion, measured by frequency of cells secreting IFN-γ by multimer analysis, intracellular cytokine staining and ELIspot.
Immune Response | baseline, weeks 1, 2, 4, 6, 8, 13, 24, 36, and 48 post-infusion
  Change in cytokine release as measured by multi-color flow cytometry
Immune Response | baseline, weeks 1, 2, 4, 6, 8, 13, 24, 36, and 48 post-infusion
  Change in polyfunctionality of HIV-1 specific CD8+ and CD4+ T-cells
Immune Response | baseline, weeks 1, 2, 4, 6, 8, 13, 24, 36, and 48 post-infusion
  Change in proportion of total and HIV-1 specific CD8+ T-cells expressing markers of immune exhaustion
Immune Response | baseline, weeks 1, 2, 4, 6, 8, 13, 24, 36, and 48 post-infusion
  Change in proportion of CD28+/CD45RA- CD8+ CTL that display effector function from baseline to post-infusion, measured by multi-color flow cytometry.
Immune Response | baseline, weeks 1, 2, 4, 6, 8, 13, 24, 36, and 48 post-infusion
  Change in antiviral activity of CD8 cells as measured by a viral inhibition assay
Immune Response | baseline, weeks 1, 2, 4, 6, 8, 13, 24, 36, and 48 post-infusion
  Change in CTL killing of resting CD4+ T cells via a novel latency clearance assay from baseline to week 13 following administration of HXTC
Virologic Measures | baseline, 4 and 13 weeks
  Change in plasma HIV-1 RNA by single copy assay (SCA)
Virologic Measures | baseline, 4 and 13 weeks
  Change in frequency of HIV-1 infection of resting CD4+ T cells using the viral outgrowth assay
Virologic Measures | baseline, 4 and 13 weeks
  Change in T-cell associated HIV-1 DNA
Virologic Measures | baseline, 4 and 13 weeks
  Change in 2LTR circles in CD4+ T cells

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gay, MD, MPH, Principal Investigator — University of North Carolina; David Margolis, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927
- [Background] Finzi D, Blankson J, Siliciano JD, Margolick JB, Chadwick K, Pierson T, Smith K, Lisziewicz J, Lori F, Flexner C, Quinn TC, Chaisson RE, Rosenberg E, Walker B, Gange S, Gallant J, Siliciano RF. Latent infection of CD4+ T cells provides a mechanism for lifelong persistence of HIV-1, even in patients on effective combination therapy. Nat Med. 1999 May;5(5):512-7. doi: 10.1038/8394. PMID 10229227
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822
- [Background] Barouch DH, Santra S, Schmitz JE, Kuroda MJ, Fu TM, Wagner W, Bilska M, Craiu A, Zheng XX, Krivulka GR, Beaudry K, Lifton MA, Nickerson CE, Trigona WL, Punt K, Freed DC, Guan L, Dubey S, Casimiro D, Simon A, Davies ME, Chastain M, Strom TB, Gelman RS, Montefiori DC, Lewis MG, Emini EA, Shiver JW, Letvin NL. Control of viremia and prevention of clinical AIDS in rhesus monkeys by cytokine-augmented DNA vaccination. Science. 2000 Oct 20;290(5491):486-92. doi: 10.1126/science.290.5491.486. PMID 11039923
- [Background] Amara RR, Villinger F, Altman JD, Lydy SL, O'Neil SP, Staprans SI, Montefiori DC, Xu Y, Herndon JG, Wyatt LS, Candido MA, Kozyr NL, Earl PL, Smith JM, Ma HL, Grimm BD, Hulsey ML, Miller J, McClure HM, McNicholl JM, Moss B, Robinson HL. Control of a mucosal challenge and prevention of AIDS by a multiprotein DNA/MVA vaccine. Science. 2001 Apr 6;292(5514):69-74. doi: 10.1126/science.1058915. PMID 11393868
- [Background] Rose NF, Marx PA, Luckay A, Nixon DF, Moretto WJ, Donahoe SM, Montefiori D, Roberts A, Buonocore L, Rose JK. An effective AIDS vaccine based on live attenuated vesicular stomatitis virus recombinants. Cell. 2001 Sep 7;106(5):539-49. doi: 10.1016/s0092-8674(01)00482-2. PMID 11551502
- [Background] Shiver JW, Fu TM, Chen L, Casimiro DR, Davies ME, Evans RK, Zhang ZQ, Simon AJ, Trigona WL, Dubey SA, Huang L, Harris VA, Long RS, Liang X, Handt L, Schleif WA, Zhu L, Freed DC, Persaud NV, Guan L, Punt KS, Tang A, Chen M, Wilson KA, Collins KB, Heidecker GJ, Fernandez VR, Perry HC, Joyce JG, Grimm KM, Cook JC, Keller PM, Kresock DS, Mach H, Troutman RD, Isopi LA, Williams DM, Xu Z, Bohannon KE, Volkin DB, Montefiori DC, Miura A, Krivulka GR, Lifton MA, Kuroda MJ, Schmitz JE, Letvin NL, Caulfield MJ, Bett AJ, Youil R, Kaslow DC, Emini EA. Replication-incompetent adenoviral vaccine vector elicits effective anti-immunodeficiency-virus immunity. Nature. 2002 Jan 17;415(6869):331-5. doi: 10.1038/415331a. PMID 11797011
- [Background] Autran B, Murphy RL, Costagliola D, Tubiana R, Clotet B, Gatell J, Staszewski S, Wincker N, Assoumou L, El-Habib R, Calvez V, Walker B, Katlama C; ORVACS Study Group. Greater viral rebound and reduced time to resume antiretroviral therapy after therapeutic immunization with the ALVAC-HIV vaccine (vCP1452). AIDS. 2008 Jul 11;22(11):1313-22. doi: 10.1097/QAD.0b013e3282fdce94. PMID 18580611
- [Background] Archin NM, Liberty AL, Kashuba AD, Choudhary SK, Kuruc JD, Crooks AM, Parker DC, Anderson EM, Kearney MF, Strain MC, Richman DD, Hudgens MG, Bosch RJ, Coffin JM, Eron JJ, Hazuda DJ, Margolis DM. Administration of vorinostat disrupts HIV-1 latency in patients on antiretroviral therapy. Nature. 2012 Jul 25;487(7408):482-5. doi: 10.1038/nature11286. PMID 22837004
- [Background] Shan L, Deng K, Shroff NS, Durand CM, Rabi SA, Yang HC, Zhang H, Margolick JB, Blankson JN, Siliciano RF. Stimulation of HIV-1-specific cytolytic T lymphocytes facilitates elimination of latent viral reservoir after virus reactivation. Immunity. 2012 Mar 23;36(3):491-501. doi: 10.1016/j.immuni.2012.01.014. Epub 2012 Mar 8. PMID 22406268
- [Background] Rosenberg ES, Altfeld M, Poon SH, Phillips MN, Wilkes BM, Eldridge RL, Robbins GK, D'Aquila RT, Goulder PJ, Walker BD. Immune control of HIV-1 after early treatment of acute infection. Nature. 2000 Sep 28;407(6803):523-6. doi: 10.1038/35035103. PMID 11029005
- [Background] Kaufmann D, Lichterfeld M, Altfeld M, al. e. Limited Durability of Immune Control following Treated Acute HIV Infection. Paper presented at: 11th Conference on Retroviruses and Opportunistic Infections; Feb 8-11, 2004; San Francisco.
- [Background] Carcelain G, Tubiana R, Samri A, Calvez V, Delaugerre C, Agut H, Katlama C, Autran B. Transient mobilization of human immunodeficiency virus (HIV)-specific CD4 T-helper cells fails to control virus rebounds during intermittent antiretroviral therapy in chronic HIV type 1 infection. J Virol. 2001 Jan;75(1):234-41. doi: 10.1128/JVI.75.1.234-241.2001. PMID 11119593
- [Background] Davey RT Jr, Bhat N, Yoder C, Chun TW, Metcalf JA, Dewar R, Natarajan V, Lempicki RA, Adelsberger JW, Miller KD, Kovacs JA, Polis MA, Walker RE, Falloon J, Masur H, Gee D, Baseler M, Dimitrov DS, Fauci AS, Lane HC. HIV-1 and T cell dynamics after interruption of highly active antiretroviral therapy (HAART) in patients with a history of sustained viral suppression. Proc Natl Acad Sci U S A. 1999 Dec 21;96(26):15109-14. doi: 10.1073/pnas.96.26.15109. PMID 10611346
- [Background] Appay V, Nixon DF, Donahoe SM, Gillespie GM, Dong T, King A, Ogg GS, Spiegel HM, Conlon C, Spina CA, Havlir DV, Richman DD, Waters A, Easterbrook P, McMichael AJ, Rowland-Jones SL. HIV-specific CD8(+) T cells produce antiviral cytokines but are impaired in cytolytic function. J Exp Med. 2000 Jul 3;192(1):63-75. doi: 10.1084/jem.192.1.63. PMID 10880527
- [Background] Janbazian L, Price DA, Canderan G, Filali-Mouhim A, Asher TE, Ambrozak DR, Scheinberg P, Boulassel MR, Routy JP, Koup RA, Douek DC, Sekaly RP, Trautmann L. Clonotype and repertoire changes drive the functional improvement of HIV-specific CD8 T cell populations under conditions of limited antigenic stimulation. J Immunol. 2012 Feb 1;188(3):1156-67. doi: 10.4049/jimmunol.1102610. Epub 2011 Dec 30. PMID 22210916
- [Background] Wherry EJ. T cell exhaustion. Nat Immunol. 2011 Jun;12(6):492-9. doi: 10.1038/ni.2035. PMID 21739672
- [Background] Wherry EJ, Blattman JN, Murali-Krishna K, van der Most R, Ahmed R. Viral persistence alters CD8 T-cell immunodominance and tissue distribution and results in distinct stages of functional impairment. J Virol. 2003 Apr;77(8):4911-27. doi: 10.1128/jvi.77.8.4911-4927.2003. PMID 12663797
- [Background] Shankar P, Russo M, Harnisch B, Patterson M, Skolnik P, Lieberman J. Impaired function of circulating HIV-specific CD8(+) T cells in chronic human immunodeficiency virus infection. Blood. 2000 Nov 1;96(9):3094-101. PMID 11049989
- [Background] Gianella S, von Wyl V, Fischer M, Niederost B, Joos B, Gunthard H, et al. Impact of early ART on proviral HIV-1 DNA and plasma viremia in acutely infected patients. In: 17th Conference on Retroviruses and Opportunistic Infections. San Francisco, CA; 2010.
- [Background] Schmid A, Gianella S, von Wyl V, Metzner KJ, Scherrer AU, Niederost B, Althaus CF, Rieder P, Grube C, Joos B, Weber R, Fischer M, Gunthard HF. Profound depletion of HIV-1 transcription in patients initiating antiretroviral therapy during acute infection. PLoS One. 2010 Oct 12;5(10):e13310. doi: 10.1371/journal.pone.0013310. PMID 20967271
- [Background] Archin NM, Cheema M, Sackman R, Sugarbaker A, Scepanski J, Kuruc J, et al. Correlation of peak and duration of viremia and resting CD4+ T-Cell infection in acute HIV infection. In: 17th Conference on Retroviruses and Opportunistic Infections, Abstract 464. San Francisco, CA; 2010.
- [Background] Hocqueloux L, Prazuck T, Avettand-Fenoel V, Lafeuillade A, Cardon B, Viard JP, Rouzioux C. Long-term immunovirologic control following antiretroviral therapy interruption in patients treated at the time of primary HIV-1 infection. AIDS. 2010 Jun 19;24(10):1598-601. doi: 10.1097/qad.0b013e32833b61ba. PMID 20549847
- [Background] Anderson JA, Archin NM, Ince W, Parker D, Wiegand A, Coffin JM, Kuruc J, Eron J, Swanstrom R, Margolis DM. Clonal sequences recovered from plasma from patients with residual HIV-1 viremia and on intensified antiretroviral therapy are identical to replicating viral RNAs recovered from circulating resting CD4+ T cells. J Virol. 2011 May;85(10):5220-3. doi: 10.1128/JVI.00284-11. Epub 2011 Mar 2. PMID 21367910
- [Background] Salazar-Gonzalez JF, Bailes E, Pham KT, Salazar MG, Guffey MB, Keele BF, Derdeyn CA, Farmer P, Hunter E, Allen S, Manigart O, Mulenga J, Anderson JA, Swanstrom R, Haynes BF, Athreya GS, Korber BT, Sharp PM, Shaw GM, Hahn BH. Deciphering human immunodeficiency virus type 1 transmission and early envelope diversification by single-genome amplification and sequencing. J Virol. 2008 Apr;82(8):3952-70. doi: 10.1128/JVI.02660-07. Epub 2008 Feb 6. PMID 18256145
- [Background] Bollard CM, Gottschalk S, Leen AM, Weiss H, Straathof KC, Carrum G, Khalil M, Wu MF, Huls MH, Chang CC, Gresik MV, Gee AP, Brenner MK, Rooney CM, Heslop HE. Complete responses of relapsed lymphoma following genetic modification of tumor-antigen presenting cells and T-lymphocyte transfer. Blood. 2007 Oct 15;110(8):2838-45. doi: 10.1182/blood-2007-05-091280. Epub 2007 Jul 3. PMID 17609424
- [Background] Hanley PJ, Shaffer DR, Cruz CR, Ku S, Tzou B, Liu H, Demmler-Harrison G, Heslop HE, Rooney CM, Gottschalk S, Bollard CM. Expansion of T cells targeting multiple antigens of cytomegalovirus, Epstein-Barr virus and adenovirus to provide broad antiviral specificity after stem cell transplantation. Cytotherapy. 2011 Sep;13(8):976-86. doi: 10.3109/14653249.2011.575356. Epub 2011 May 4. PMID 21539497
- [Background] Lieberman J, Skolnik PR, Parkerson GR 3rd, Fabry JA, Landry B, Bethel J, Kagan J. Safety of autologous, ex vivo-expanded human immunodeficiency virus (HIV)-specific cytotoxic T-lymphocyte infusion in HIV-infected patients. Blood. 1997 Sep 15;90(6):2196-206. PMID 9310470
- [Background] Chapuis AG, Casper C, Kuntz S, Zhu J, Tjernlund A, Diem K, Turtle CJ, Cigal ML, Velez R, Riddell S, Corey L, Greenberg PD. HIV-specific CD8+ T cells from HIV+ individuals receiving HAART can be expanded ex vivo to augment systemic and mucosal immunity in vivo. Blood. 2011 May 19;117(20):5391-402. doi: 10.1182/blood-2010-11-320226. Epub 2011 Mar 21. PMID 21422474
- [Background] Tan R, Xu X, Ogg GS, Hansasuta P, Dong T, Rostron T, Luzzi G, Conlon CP, Screaton GR, McMichael AJ, Rowland-Jones S. Rapid death of adoptively transferred T cells in acquired immunodeficiency syndrome. Blood. 1999 Mar 1;93(5):1506-10. PMID 10029578
- [Background] Brodie SJ, Lewinsohn DA, Patterson BK, Jiyamapa D, Krieger J, Corey L, Greenberg PD, Riddell SR. In vivo migration and function of transferred HIV-1-specific cytotoxic T cells. Nat Med. 1999 Jan;5(1):34-41. doi: 10.1038/4716. PMID 9883837
- [Background] Whiteside TL, Elder EM, Moody D, Armstrong J, Ho M, Rinaldo C, Huang X, Torpey D, Gupta P, McMahon D, et al. Generation and characterization of ex vivo propagated autologous CD8+ cells used for adoptive immunotherapy of patients infected with human immunodeficiency virus. Blood. 1993 Apr 15;81(8):2085-92. PMID 8471767
- [Background] Ho M, Armstrong J, McMahon D, Pazin G, Huang XL, Rinaldo C, Whiteside T, Tripoli C, Levine G, Moody D, et al. A phase 1 study of adoptive transfer of autologous CD8+ T lymphocytes in patients with acquired immunodeficiency syndrome (AIDS)-related complex or AIDS. Blood. 1993 Apr 15;81(8):2093-101. PMID 8471768
- [Background] Torpey D 3rd, Huang XL, Armstrong J, Ho M, Whiteside T, McMahon D, Pazin G, Heberman R, Gupta P, Tripoli C, et al. Effects of adoptive immunotherapy with autologous CD8+ T lymphocytes on immunologic parameters: lymphocyte subsets and cytotoxic activity. Clin Immunol Immunopathol. 1993 Sep;68(3):263-72. doi: 10.1006/clin.1993.1127. PMID 8370181
- [Background] Koenig S, Conley AJ, Brewah YA, Jones GM, Leath S, Boots LJ, Davey V, Pantaleo G, Demarest JF, Carter C, et al. Transfer of HIV-1-specific cytotoxic T lymphocytes to an AIDS patient leads to selection for mutant HIV variants and subsequent disease progression. Nat Med. 1995 Apr;1(4):330-6. doi: 10.1038/nm0495-330. PMID 7585062
- [Background] Saavedra S, Sanz GF, Jarque I, Moscardo F, Jimenez C, Lorenzo I, Martin G, Martinez J, De La Rubia J, Andreu R, Molla S, Llopis I, Fernandez MJ, Salavert M, Acosta B, Gobernado M, Sanz MA. Early infections in adult patients undergoing unrelated donor cord blood transplantation. Bone Marrow Transplant. 2002 Dec;30(12):937-43. doi: 10.1038/sj.bmt.1703764. PMID 12476288
- [Background] Bollard CM, Gottschalk S, Torrano V, Diouf O, Ku S, Hazrat Y, Carrum G, Ramos C, Fayad L, Shpall EJ, Pro B, Liu H, Wu MF, Lee D, Sheehan AM, Zu Y, Gee AP, Brenner MK, Heslop HE, Rooney CM. Sustained complete responses in patients with lymphoma receiving autologous cytotoxic T lymphocytes targeting Epstein-Barr virus latent membrane proteins. J Clin Oncol. 2014 Mar 10;32(8):798-808. doi: 10.1200/JCO.2013.51.5304. Epub 2013 Dec 16. PMID 24344220
- [Background] Rosenberg ES, Billingsley JM, Caliendo AM, Boswell SL, Sax PE, Kalams SA, Walker BD. Vigorous HIV-1-specific CD4+ T cell responses associated with control of viremia. Science. 1997 Nov 21;278(5342):1447-50. doi: 10.1126/science.278.5342.1447. PMID 9367954
- [Background] Volberding P, Demeter L, Bosch RJ, Aga E, Pettinelli C, Hirsch M, Vogler M, Martinez A, Little S, Connick E; ACTG 371 Team. Antiretroviral therapy in acute and recent HIV infection: a prospective multicenter stratified trial of intentionally interrupted treatment. AIDS. 2009 Sep 24;23(15):1987-95. doi: 10.1097/QAD.0b013e32832eb285. PMID 19696651
- [Background] Hecht FM, Wang L, Collier A, Little S, Markowitz M, Margolick J, Kilby JM, Daar E, Conway B, Holte S; AIEDRP Network. A multicenter observational study of the potential benefits of initiating combination antiretroviral therapy during acute HIV infection. J Infect Dis. 2006 Sep 15;194(6):725-33. doi: 10.1086/506616. Epub 2006 Aug 15. PMID 16941337
- [Background] Ortiz GM, Nixon DF, Trkola A, Binley J, Jin X, Bonhoeffer S, Kuebler PJ, Donahoe SM, Demoitie MA, Kakimoto WM, Ketas T, Clas B, Heymann JJ, Zhang L, Cao Y, Hurley A, Moore JP, Ho DD, Markowitz M. HIV-1-specific immune responses in subjects who temporarily contain virus replication after discontinuation of highly active antiretroviral therapy. J Clin Invest. 1999 Sep;104(6):R13-8. doi: 10.1172/JCI7371. PMID 10491418
- [Background] Steingrover R, Pogany K, Fernandez Garcia E, Jurriaans S, Brinkman K, Schuitemaker H, Miedema F, Lange JM, Prins JM. HIV-1 viral rebound dynamics after a single treatment interruption depends on time of initiation of highly active antiretroviral therapy. AIDS. 2008 Aug 20;22(13):1583-8. doi: 10.1097/QAD.0b013e328305bd77. PMID 18670217
- [Background] Bongiovanni M, Casana M, Tincati C, d'Arminio Monforte A. Treatment interruptions in HIV-infected subjects. J Antimicrob Chemother. 2006 Sep;58(3):502-5. doi: 10.1093/jac/dkl268. Epub 2006 Jul 1. PMID 16816398
- [Background] Rosenberg ZF, Fauci AS. Immunopathogenic mechanisms of HIV infection: cytokine induction of HIV expression. Immunol Today. 1990 May;11(5):176-80. doi: 10.1016/0167-5699(90)90070-p. PMID 2186752
- [Background] Pilcher CD, Eron JJ Jr, Galvin S, Gay C, Cohen MS. Acute HIV revisited: new opportunities for treatment and prevention. J Clin Invest. 2004 Apr;113(7):937-45. doi: 10.1172/JCI21540. PMID 15057296
- [Background] Pires A, Hardy G, Gazzard B, Gotch F, Imami N. Initiation of antiretroviral therapy during recent HIV-1 infection results in lower residual viral reservoirs. J Acquir Immune Defic Syndr. 2004 Jul 1;36(3):783-90. doi: 10.1097/00126334-200407010-00004. PMID 15213561
- [Background] Ramratnam B, Ribeiro R, He T, Chung C, Simon V, Vanderhoeven J, Hurley A, Zhang L, Perelson AS, Ho DD, Markowitz M. Intensification of antiretroviral therapy accelerates the decay of the HIV-1 latent reservoir and decreases, but does not eliminate, ongoing virus replication. J Acquir Immune Defic Syndr. 2004 Jan 1;35(1):33-7. doi: 10.1097/00126334-200401010-00004. PMID 14707789
- [Background] Chamberland A, Sylla M, Boulassel MR, Baril JG, Cote P, Thomas R, Trottier B, Rouleau D, Routy JP, Tremblay C; Investigators of the Primary HIV-Infection Cohort of Montreal. Effect of antiretroviral therapy on HIV-1 genetic evolution during acute infection. Int J STD AIDS. 2011 Mar;22(3):146-50. doi: 10.1258/ijsa.2010.010292. PMID 21464451
- [Background] Gay CL, Mayo AJ, Mfalila CK, Chu H, Barry AC, Kuruc JD, McGee KS, Kerkau M, Sebastian J, Fiscus SA, Margolis DM, Hicks CB, Ferrari G, Eron JJ; Duke-UNC Acute HIV Infection Consortium. Efficacy of NNRTI-based antiretroviral therapy initiated during acute HIV infection. AIDS. 2011 Apr 24;25(7):941-9. doi: 10.1097/QAD.0b013e3283463c07. PMID 21487250
- [Background] Gay C, Dibben O, Anderson JA, Stacey A, Mayo AJ, Norris PJ, Kuruc JD, Salazar-Gonzalez JF, Li H, Keele BF, Hicks C, Margolis D, Ferrari G, Haynes B, Swanstrom R, Shaw GM, Hahn BH, Eron JJ, Borrow P, Cohen MS. Cross-sectional detection of acute HIV infection: timing of transmission, inflammation and antiretroviral therapy. PLoS One. 2011 May 10;6(5):e19617. doi: 10.1371/journal.pone.0019617. PMID 21573003
- [Background] Keedy KS, Archin NM, Gates AT, Espeseth A, Hazuda DJ, Margolis DM. A limited group of class I histone deacetylases acts to repress human immunodeficiency virus type 1 expression. J Virol. 2009 May;83(10):4749-56. doi: 10.1128/JVI.02585-08. Epub 2009 Mar 11. PMID 19279091
- [Background] Palmer S, Wiegand AP, Maldarelli F, Bazmi H, Mican JM, Polis M, Dewar RL, Planta A, Liu S, Metcalf JA, Mellors JW, Coffin JM. New real-time reverse transcriptase-initiated PCR assay with single-copy sensitivity for human immunodeficiency virus type 1 RNA in plasma. J Clin Microbiol. 2003 Oct;41(10):4531-6. doi: 10.1128/JCM.41.10.4531-4536.2003. PMID 14532178
- [Background] Archin NM, Eron JJ, Palmer S, Hartmann-Duff A, Martinson JA, Wiegand A, Bandarenko N, Schmitz JL, Bosch RJ, Landay AL, Coffin JM, Margolis DM. Valproic acid without intensified antiviral therapy has limited impact on persistent HIV infection of resting CD4+ T cells. AIDS. 2008 Jun 19;22(10):1131-5. doi: 10.1097/QAD.0b013e3282fd6df4. PMID 18525258
- [Background] Gandhi RT, Zheng L, Bosch RJ, Chan ES, Margolis DM, Read S, Kallungal B, Palmer S, Medvik K, Lederman MM, Alatrakchi N, Jacobson JM, Wiegand A, Kearney M, Coffin JM, Mellors JW, Eron JJ; AIDS Clinical Trials Group A5244 team. The effect of raltegravir intensification on low-level residual viremia in HIV-infected patients on antiretroviral therapy: a randomized controlled trial. PLoS Med. 2010 Aug 10;7(8):e1000321. doi: 10.1371/journal.pmed.1000321. PMID 20711481
- [Derived] Sung JA, Patel S, Clohosey ML, Roesch L, Tripic T, Kuruc JD, Archin N, Hanley PJ, Cruz CR, Goonetilleke N, Eron JJ, Rooney CM, Gay CL, Bollard CM, Margolis DM. HIV-Specific, Ex Vivo Expanded T Cell Therapy: Feasibility, Safety, and Efficacy in ART-Suppressed HIV-Infected Individuals. Mol Ther. 2018 Oct 3;26(10):2496-2506. doi: 10.1016/j.ymthe.2018.08.015. Epub 2018 Sep 21. PMID 30249388
- See also: University of North Carolina — http://www.unc.edu